CLINICAL TRIAL: NCT05877027
Title: Comparison of Commonly Used Treatment Approaches in the Treatment of Gonarthrosis: Platelet-Rich Plasma, Topical Diclofenac, and Exercise
Brief Title: Exercise vs. Topical Diclofenac vs. PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sezen Karaborklu Argut, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4370438302
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Gonarthrosis
Keywords: Physiotherapy; Non-steroidal anti-inflammatory drugs; Intraarticular Injection; Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Exercise; Diclofenac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator administering the treatment and the investigator performing the evaluations will be different. The evaluator will not know about the interventions that the participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group 1 (Active Comparator): The patients in the Exercise group will be treated with a structured exercise program. The exercises will be applied by the research physiotherapist for 6 weeks, 2 days a week. Each training session is planned to last approximately 30 minutes.
  Interventions: Other: Exercise
- Intervention Group 2 (Active Comparator): The patients in the topical agent group were prescribed by the orthopedist. they will use the topical agent. Diclofenac in gel form was chosen as a topical agent in the light of the literature. In this context, patients in both groups will apply the topical agent around the knee joint 4 days a week, 2 times a day (every 12 hours) in the morning and evening for 6 weeks.
  Interventions: Other: Topical Diclofenac
- Intervention Group 3 (Active Comparator): The PRP procedure with the same characteristics will be used in the treatment of patients in the PRP group. The PRP application will be prepared by the orthopedics and traumatology specialist physician in the research team, using the kits provided within the scope of the project. In order to collect venous blood for the PRP production procedure, gamma sterile vacuum tubes and blood collection set in special kits without the risk of contamination will be used. A total of 3 doses will be administered to the patients, with a one-week interval between doses.
  Interventions: Other: Platelet-Rich-Plasma (PRP)

INTERVENTIONS:
Other: Exercise — The first 3 weeks of the exercise program will include range of motion exercises, isometric and isotonic strengthening exercises for the muscles around the knee and hip, and stretching exercises. In the following 3 weeks, resistance strengthening exercises and closed kinetic chain exercises will be added to the program.
  Arms: Intervention Group 1
Other: Topical Diclofenac — They will apply it around the knee joint 4 days a week, 2 times a day (every 12 hours), morning and evening for 6 weeks.
  Arms: Intervention Group 2
Other: Platelet-Rich-Plasma (PRP) — 8 ml of blood will be taken from each patient in tubes containing 0.9 ml of 3.2% sodium citrate. Swing-out rotor (open-swing type) will be placed in the centrifuge with the tubes facing each other. After centrifugation, 2.5 cc of PRP product will be collected from each tube and the resulting PRP will be administered to patients by injection under sterile conditions.
  Arms: Intervention Group 3

SUMMARY:
Osteoarthritis, the most common type of arthritis, is a chronic and degenerative joint disease. It has been reported to affect more than 300 million adults and elderly individuals worldwide. The joint most commonly affected by osteoarthritis is the knee joint and this condition is called gonarthrosis.

The goal of treatment is to reduce symptoms and ultimately slow the progression of the disease with various treatment options throughout the course of the disease.Current clinical studies prepared by the working groups of the International Osteoarthritis Research Society (OARSI) and the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO) According to the guidelines, treatment typically includes physiotherapy interventions with the use of non-steroidal anti-inflammatory drugs (NSAIDs) and analgesics, including intra-articular injections of corticosteroids. Exercise-oriented physiotherapy is one of the main approaches for the conservative treatment of gonarthrosis. The curative clinical effect of exercise therapy on pain and functional disability in gonarthrosis is important.

The use of PRP in the treatment of gonarthrosis is based on the ability of platelets to release biologically active proteins and promote tissue healing. Since the cartilage tissue mainly affected in gonarthrosis has low healing potential, this feature of platelets becomes more important for the target tissue. Existing studies show that PRP is superior to hyaluronic acid in intermediate and initial gonarthrosis; on the other hand, less satisfactory results are reported in severe gonarthrosis, similar to viscosupplementation.

Topically or orally administered NSAIDs form the backbone of pharmacological treatment in gonarthrosis.

It is seen that both exercise, PRP and topical NSAID agents are among the recommendations in the treatment of gonarthrosis. However, there is insufficient evidence regarding the superiority and therapeutic efficacy of these three treatment approaches. The aim of this study is to determine the effectiveness of "exercise", "PRP" and "NSAID-specific topical agents" in the treatment of patients with gonarthrosis; pain, function, quality of life, and patient satisfaction.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with gonarthritis will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into tree groups. Study groups will be as follows: a) exercise, b) topical diclofenac, c) platalet-rich-plasma (PRP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gonarthrosis according to the criteria of the American Society of Rheumatology (ACR)
* Stage 2 or 3 according to Kellgren Lawrence radiological staging criteria,
* Those between the ages of 40 and 65,
* Body mass index below 30 kg/m2,
* Pain intensity defined by the patient in the last 3 months is at least 3 out of 10 according to NPRS,
* Patients who do not have any barriers to being included in the exercise program

Exclusion Criteria:

* Being in stage 4 according to Kellgren Lawrence radiological staging criteria,
* Hemoglobin level <11.5 g/dL
* Platelet level <100,000/μL
* Thrombocytopenia, coagulopathy, crystal arthropathy, hemophilia or hematological malignancy,
* Presence of active infection or tumor,
* Chronic antiaggregant use or taking immunosuppressive therapy,
* Pregnancy or lactation,
* Viscosupplementation or steroid injection in the related knee in the last 3 months, or using systemic steroids,
* To have received a physiotherapy program for the relevant knee in the last 3 months,
* Having a valgus or varus deformity greater than 15°,
* Presence of neurological diseases and/or deformity leading to lower extremity muscle weakness
* Having serious systemic and cardiovascular diseases that interfere with exercise

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
Change of Pain via Numeric Pain Rating Scale | change from baseline pain at 6 months
  On this scale, "0" indicates the absence of pain, and "10" indicates the most severe pain imaginable. Patients will be asked to rate the severity of their knee pain with a number between 0 and 10 using this scale. The minimum clinically significant difference value (MCID) of this valid and reliable pain scale is 1.74 points.

SECONDARY OUTCOMES:
WOMAC | 4 times for 24 weeks
  WOMAC assesses the level of difficulty, pain and joint stiffness experienced by the patients during their physical functions. WOMAC score is a 5-point Likert-type scale, high scores indicate poor status and consist of a total of 24 questions.
40 meters fast walking test | 4 times for 24 weeks
  For 40mHYT, patients will be asked to walk as fast as possible on a flat and hard surface, on a 10-meter marked walking path. Walking time will be measured in seconds with a stopwatch. The test will be repeated three times and the arithmetic mean of these measurements will be recorded as the result value. Considering the age range of the patients, it was planned to allow a one-minute rest period between retests.
Stepping Test | 4 times for 24 weeks
  Patients will be asked to climb 10 pre-marked 20 cm high steps as quickly as possible on a standard ladder. The test time will be measured in seconds with a stopwatch. The test will be repeated 3 times and the average value will be recorded in seconds. Similarly, in this evaluation, patients were given a one-minute rest period between 3 repetitions of the test.
Joint Range of Motion Evaluation | 4 times for 24 weeks
  During the assessments, three repeat measurements will be made using an electronic goniometer. For goniometric measurement, the pivot point will be placed on the lateral condyle of the femur. The fixed arm will be held parallel to the lateral midline of the femur. The movable arm will follow the movement of the fibula.
Health-Related Quality of Life Short Form-12 Scale (SF-12) | 4 times for 24 weeks
  SF-12 is the abbreviated version of the Short Form-36 (SF-36) Quality of Life Scale and is frequently preferred for ease of use. It has 2 components, physical and mental, scored between 0 and 50. A high score from the score indicates health-related well-being and increased quality of life, while a decrease indicates worsening.
Global Rating of Change Scale-GRC | 4 times for 24 weeks
  It will be used to evaluate patient satisfaction. It is designed to determine the amount of improvement or worsening of the patient over time. In our study, GRC consisting of 5 levels between -2 and +2 value ranges (-2: I am much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better) was preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Karabörklü Argut, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Safiri S, Kolahi AA, Smith E, Hill C, Bettampadi D, Mansournia MA, Hoy D, Ashrafi-Asgarabad A, Sepidarkish M, Almasi-Hashiani A, Collins G, Kaufman J, Qorbani M, Moradi-Lakeh M, Woolf AD, Guillemin F, March L, Cross M. Global, regional and national burden of osteoarthritis 1990-2017: a systematic analysis of the Global Burden of Disease Study 2017. Ann Rheum Dis. 2020 Jun;79(6):819-828. doi: 10.1136/annrheumdis-2019-216515. Epub 2020 May 12. PMID 32398285
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] Bruyere O, Honvo G, Veronese N, Arden NK, Branco J, Curtis EM, Al-Daghri NM, Herrero-Beaumont G, Martel-Pelletier J, Pelletier JP, Rannou F, Rizzoli R, Roth R, Uebelhart D, Cooper C, Reginster JY. An updated algorithm recommendation for the management of knee osteoarthritis from the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Semin Arthritis Rheum. 2019 Dec;49(3):337-350. doi: 10.1016/j.semarthrit.2019.04.008. Epub 2019 Apr 30. PMID 31126594
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Gregori D, Giacovelli G, Minto C, Barbetta B, Gualtieri F, Azzolina D, Vaghi P, Rovati LC. Association of Pharmacological Treatments With Long-term Pain Control in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. JAMA. 2018 Dec 25;320(24):2564-2579. doi: 10.1001/jama.2018.19319. PMID 30575881
- [Background] Arden NK, Perry TA, Bannuru RR, Bruyere O, Cooper C, Haugen IK, Hochberg MC, McAlindon TE, Mobasheri A, Reginster JY. Non-surgical management of knee osteoarthritis: comparison of ESCEO and OARSI 2019 guidelines. Nat Rev Rheumatol. 2021 Jan;17(1):59-66. doi: 10.1038/s41584-020-00523-9. Epub 2020 Oct 28. PMID 33116279
- [Background] van Doormaal MCM, Meerhoff GA, Vliet Vlieland TPM, Peter WF. A clinical practice guideline for physical therapy in patients with hip or knee osteoarthritis. Musculoskeletal Care. 2020 Dec;18(4):575-595. doi: 10.1002/msc.1492. Epub 2020 Jul 9. PMID 32643252
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142